CLINICAL TRIAL: NCT04756427
Title: Sodium Citrate 4% Locking Solution for Children Requiring Home Parenteral Nutrition
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Subject recruitment was challenging
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00264457
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Results first posted 2024-09-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: CLABSI - Central Line Associated Bloodstream Infection
Keywords: pediatric; home parenteral nutrition; intestinal failure
MeSH Terms: conditions — Intestinal Failure | interventions — Sodium Citrate

STUDY DESIGN:
Intervention Model Description: Prospective cohort after intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Sodium citrate 4% (Experimental): All enrolled participants will received the daily sodium citrate 4% locking solution for CLABSI prophylaxis intervention and be observed prospectively for adverse events
  Interventions: Drug: Sodium Citrate 4% Inj Syringe 3Ml

INTERVENTIONS:
Drug: Sodium Citrate 4% Inj Syringe 3Ml — 3 ml of sodium citrate 4% locking solution instilled into the central catheter daily during the period that parenteral nutrition is not infusing, and will be withdrawn and disposed of prior to resuming infusion of parenteral nutrition
  Other Names: ANDA BA125608 / Sodium Citrate 4% w/v Anticoagulant Solution USP

SUMMARY:
This study an open label prospective observational cohort study to evaluate the safety and efficacy of sodium citrate 4% locking solution in preventing central line associated blood stream infection in children requiring long term central venous catheters for home parenteral nutrition. Sodium citrate 4% is FDA-approved for dialysis catheters, but has not been formally evaluated for use in tunneled catheters for parenteral nutrition. The rate of central line-associated bloodstream infection (CLABSI) and other potential adverse events will be monitored for 12 months, with the option to remain in the study for a longer period of time.

DETAILED DESCRIPTION:
In this prospective observational cohort study of pediatric patients requiring home parenteral nutrition for intestinal failure, participants will be enrolled from the pediatric intestinal rehabilitation clinic, and data collection will be obtained from the electronic medical record. Participant will receive daily sodium citrate 4% catheter locking solution for CLABSI prophylaxis, instead of heparin locks. Participants will be monitored for 12 months for adverse events, including CLABSI. Participants will have the same routine laboratory schedule and monthly outpatient follow up. After 12 months, participants will be given the option to continue to use sodium citrate 4% locks after the initial study period if no serious adverse events have occurred. The investigators anticipate enrolling 10-15 participants per year and anticipate enrollment to continue for 3-5 years.

Sodium citrate locks: 3 ml vials of locking solution will be prepared by the infusion pharmacy using commercially available 4% sodium citrate IV fluid (available in 500 ml bags). The sodium citrate locks will be instilled into the central catheter daily during the period that parenteral nutrition is not infusing, and will be withdrawn and disposed of prior to resuming infusion of parenteral nutrition. If subjects are hospitalized, sodium citrate locks will be temporarily held during the duration of the inpatient stay, and will be resumed once the participant is discharged home.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (<18 years) and adult patients (up to 21 years still in our clinic)
* requiring long-term (>3 months) home parenteral nutrition due to intestinal failure/short bowel syndrome
* has had at least one central line-associated blood stream infection

Exclusion Criteria:

* known cardiac arrhythmias
* hypersensitivity to citrate
* pregnancy
* receiving continuous parenteral nutrition (infusing over 24 hours)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darla Shores, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
de-identified data (demographics, outcomes) may be shared upon request

REFERENCES:
- [Background] Passero BA, Zappone P, Lee HE, Novak C, Maceira EL, Naber M. Citrate versus heparin for apheresis catheter locks: an efficacy analysis. J Clin Apher. 2015 Feb;30(1):22-7. doi: 10.1002/jca.21346. Epub 2014 Aug 13. PMID 25132635
- [Background] Grudzinski L, Quinan P, Kwok S, Pierratos A. Sodium citrate 4% locking solution for central venous dialysis catheters--an effective, more cost-efficient alternative to heparin. Nephrol Dial Transplant. 2007 Feb;22(2):471-6. doi: 10.1093/ndt/gfl606. Epub 2006 Oct 25. PMID 17065193
- [Background] Pittiruti M, Bertoglio S, Scoppettuolo G, Biffi R, Lamperti M, Dal Molin A, Panocchia N, Petrosillo N, Venditti M, Rigo C, DeLutio E. Evidence-based criteria for the choice and the clinical use of the most appropriate lock solutions for central venous catheters (excluding dialysis catheters): a GAVeCeLT consensus. J Vasc Access. 2016 Nov 2;17(6):453-464. doi: 10.5301/jva.5000576. Epub 2016 Aug 1. PMID 27516141
- [Background] Weijmer MC, Debets-Ossenkopp YJ, Van De Vondervoort FJ, ter Wee PM. Superior antimicrobial activity of trisodium citrate over heparin for catheter locking. Nephrol Dial Transplant. 2002 Dec;17(12):2189-95. doi: 10.1093/ndt/17.12.2189. PMID 12454232
- [Background] Michaud D, Komant T, Pfefferle P. Four percent trisodium citrate as an alternative anticoagulant for maintaining patency of central venous hemodialysis catheters: case report and discussion. Am J Crit Care. 2001 Sep;10(5):351-4. No abstract available. PMID 11548568
- [Background] Battistella M, Vercaigne LM, Cote D, Lok CE. Antibiotic lock: in vitro stability of gentamicin and sodium citrate stored in dialysis catheters at 37 degrees C. Hemodial Int. 2010 Jul;14(3):322-6. doi: 10.1111/j.1542-4758.2010.00440.x. Epub 2009 Mar 24. PMID 20345391
- [Background] Grudzinski A, Agarwal A, Bhatnagar N, Nesrallah G. Benefits and harms of citrate locking solutions for hemodialysis catheters: a systematic review and meta-analysis. Can J Kidney Health Dis. 2015 Apr 2;2:13. doi: 10.1186/s40697-015-0040-2. eCollection 2015. PMID 25926995

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only 1 participant was enrolled in this study. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Period: Overall Study
Arm/Group | Sodium Citrate 4%
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Only 1 participant was enrolled in this study. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Arm/Group | Sodium Citrate 4%
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Central Line-associated Bloodstream Infection (CLABSI) Rate
Description: Frequency of fever with positive central line blood culture events per central line days.
Time Frame: 12 months
Population: as for baseline characteristics
Arm/Group | Sodium Citrate 4%
Number analyzed (Participants) | 0

2. Secondary Outcome: Central Venous Catheter Thrombus Rate
Description: Central line thrombus events requiring anti-coagulation treatment per central line days.
Time Frame: 12 months
Population: as for baseline characteristics
Arm/Group | Sodium Citrate 4%
Number analyzed (Participants) | 0

3. Secondary Outcome: Central Line Removal Rate
Description: Central line removal events (infection or other dysfunction) per central line days.
Time Frame: 12 months
Population: as for baseline characteristics
Arm/Group | Sodium Citrate 4%
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Serious Adverse Events
Description: Serious adverse events will be assessed with number of hospitalizations for any reason.
Time Frame: 12 months
Population: as for baseline characteristics
Arm/Group | Sodium Citrate 4%
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Only 1 participant was enrolled in this study. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Description: Only 1 participant was enrolled in this study. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Arm/Group | Sodium Citrate 4%
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/27/NCT04756427/Prot_SAP_000.pdf